CLINICAL TRIAL: NCT00288574
Title: Fluoxetine After Weight Restoration in Anorexia Nervosa
Brief Title: Fluoxetine to Prevent Relapse and Enhance Psychological Recovery in Women With Anorexia Nervosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #4703R; R01MH060271 (NIH); R01MH060336 (NIH); DSIR AT-P
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Anorexia Nervosa; Eating Disorders
Keywords: Depression
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- fluoxetine (Experimental): fluoxetine up to 80 mg per day
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine
  Arms: fluoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of fluoxetine versus placebo in reducing the rate of relapse of anorexia nervosa (AN) and enhancing the psychosocial and behavioral recovery of people who have been treated for AN.

DETAILED DESCRIPTION:
Anorexia nervosa (AN), a type of eating disorder, is a serious psychiatric illness that is characterized by an extreme loss of appetite. People with AN view themselves as overweight and cannot bring themselves to eat, even though most are dangerously thin. Signs of the disorder include unusual eating habits, such as avoiding food and meals, picking out a few foods and eating them in small quantities, or carefully weighing and portioning food. Some people with AN fully recover after a single episode, some have a fluctuating pattern of weight gain and relapse, and others experience a chronic course of illness over many years. Effective drugs to treat the disorder are lacking. In addition, most past research has examined the effect of medications during the initial phase of treatment, a time when AN patients may not respond to medication because of the acute effects of starvation. Fluoxetine is a selective serotonin reuptake inhibitor (SSRI) that is commonly used to treat depression. This study will evaluate the effectiveness of fluoxetine versus placebo in reducing the rate of relapse of AN and enhancing the psychosocial and behavioral recovery of women who have already been treated for AN.

Participants in this double-blind study will be recruited immediately following completion of a treatment program for AN, in which they maintained a body mass index (BMI) of at least 19 kg/m2 for two weeks. Upon study entry, participants will be randomly assigned to receive either fluoxetine or placebo for 12 months. Participants will begin receiving medication one week prior to discharge from the hospital in which they received care for AN. Medication doses will be increased up to a target dose of 60 mg per day, and will not exceed 80 mg per day. Participants will receive 50 sessions of cognitive-behavioral therapy, lasting approximately 45 minutes each and occurring twice weekly for the first month following discharge from the hospital. After the first month, therapy sessions will occur once weekly until Month 9 and then every other week until Month 12. Participants will also report to the study site to meet with a psychiatrist once a week for the first month following discharge and then every other week for the remainder of the study. General medical status, evidence of AN relapse, medication dose, and side effects will be assessed at these visits. Upon completing treatment, follow-up telephone calls will occur at Months 15 and 21, and follow-up visits will be held at Months 18 and 24. Psychopathology associated with AN, including concern with weight and shape, depressive symptoms, anxiety, and obsessive behavior, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for anorexia nervosa (except the requirement for amenorrhea)
* Successfully completed treatment at one of the study sites in an inpatient or day-program setting immediately prior to study entry (BMI remained at least 19 kg/m2 for two weeks)

Exclusion Criteria:

* Currently taking any medications other than occasional lorazepam or zopiclone for anxiety or sleep disturbance
* Previous serious adverse reactions to fluoxetine (e.g., allergy)
* Currently at risk for suicide
* Any medical condition requiring treatment with other psychotropic medication (except the occasional use of anti-anxiety medication)
* Pregnant
* Any serious medical illness besides the eating disorder
* History of continuous illness (at a low weight with no periods of remission or return to normal functioning for more than 15 years)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2000-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Timothy Walsh, MD, Principal Investigator — New York State Psychiatric Institute/Columbia University Medical Center; Allan Kaplan, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- New York State Psychiatric Institute/Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Walsh BT, Kaplan AS, Attia E, Olmsted M, Parides M, Carter JC, Pike KM, Devlin MJ, Woodside B, Roberto CA, Rockert W. Fluoxetine after weight restoration in anorexia nervosa: a randomized controlled trial. JAMA. 2006 Jun 14;295(22):2605-12. doi: 10.1001/jama.295.22.2605. PMID 16772623

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine: fluoxetine up to 80 mg per day
  Fluoxetine
- Placebo: Placebo group
Period: Overall Study
Arm/Group | Fluoxetine | Placebo
Started | 49 | 44
Completed | 49 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 49 | 44 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 44 | 93
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (4.46) | 24.2 (4.52) | 23 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 44 | 93
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 19 | 45
  Canada | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Remaining in Study at 1 Year
Description: The primary outcome measure was the proportion of patients with AN successfully completing 1 year of treatment and maintaining > 85% Ideal Body Weight.
Time Frame: 12 months
Measure: Number; unit: proportion of participants
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
proportion of participants | 0.265 | 0.315
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; The proportion of patients successfully completing the trial in the fluoxetine and placebo groups was compared using the chi-squared statistic; Test type: Superiority; p = 0.57, Chi-squared

2. Secondary Outcome: Change in Weight Per Month During Treatment
Time Frame: 12 months
Measure: Mean (Standard Error); unit: kg per month
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
kg per month | -1.94 (0.51) | -2.14 (0.33)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment in body weight, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.75, Mixed Models Analysis — Reported p values of secondary measures were not corrected for multiple comparisons. The Bonferroni corrected level of significance is <0.005

3. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With Beck Anxiety Inventory (BAI)
Description: The Beck Anxiety Inventory is a 21 question self-report measure of anxiety symptoms during the past week. Possible scores range from 0 - 63, with higher scores indicating more severe symptoms. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: placebo to match fluoxetine
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | -0.70 (0.12) | -0.22 (0.13)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment of BDI in fluoxetine versus placebo groups; Test type: Superiority; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With Beck Depression Inventory (BDI)
Description: The Beck Depression Inventory-II is a 21 question self-report measure of depressive symptoms. Possible scores range from 0 - 63, with higher scores indicating more severe symptoms.Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | 0.12 (0.25) | 0.20 (0.17)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment in BDI, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.79, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Rosenberg Self-Esteem Scale (RSES).
Description: The RSES is a 10 item self-report measure of self-esteem. Possible scores range from 0 - 30, with lower scores indicating more severe symptoms. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | 0.12 (0.08) | 0.07 (0.08)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment in RSES, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.69, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q).
Description: The Q-LES-Q is a 93 item self-report measure of enjoyment and satisfaction experienced by individuals in various areas of daily functioning. Each of the 93 items is scored on a five-point scale, and the total score is converted to a percentage of the maximum score possible. The range is therefore from 0 to 100, with a higher score indicating greater enjoyment or satisfaction. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: percentage of maximum possible score
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
percentage of maximum possible score | 0.23 (0.23) | 0.31 (0.18)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment in Q-LES-Q, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.78, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Eating Disorders Inventory (EDI), Drive for Thinness Subscale.
Description: The EDI is a 64 item self-report measure of psychological and behavioral characteristics of eating disorders. The Drive for Thinness subscale is comprised of seven items indicating excessive concern with dieting, preoccupation with weight and entrenchment in an extreme pursuit of thinness. Possible scores range from 0 to 21, with higher scores indicating greater Drive for Thinness. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | -0.24 (0.09) | -0.81 (0.09)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment in Drive for Thinness subscale, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.19, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

8. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Eating Disorders Inventory (EDI), Bulimia Subscale.
Description: The EDI is a 64 item self-report measure of psychological and behavioral characteristics of eating disorders. The Bulimia subscale is comprised of seven items indicating the tendency towards episodes of uncontrollable overeating (binge eating). Possible scores range from 0 to 21, with higher scores indicating greater tendency. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | -0.11 (0.07) | 0.035 (0.08)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment in Bulimia subscale, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.46, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

9. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Eating Disorders Inventory (EDI), Body Dissatisfaction Subscale.
Description: The EDI is a 64 item self-report measure of psychological and behavioral characteristics of eating disorders. The Body Dissatisfaction subscale is comprised of nine items indicating the belief that parts of the body are too large. Possible scores range from 0 to 27, with higher scores indicating greater dissatisfaction. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | -0.24 (0.09) | -0.26 (0.09)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment on Body Dissatisfaction subscale, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.86, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

10. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Eating Disorders Inventory (EDI), Perfectionism Subscale.
Description: The EDI is a 64 item self-report measure of psychological and behavioral characteristics of eating disorders. The Perfectionism subscale is comprised of six items Indicating excessive personal expectations for superior achievement. Possible scores range from 0 to 18, with higher scores indicating greater expectations. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | -0.037 (0.03) | 0.05 (0.06)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment on Perfectionism subscale, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.25, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

11. Secondary Outcome: Change Per Month in Psychological Symptoms During Treatment, Assessed With the Yale Brown Cornell Obsessive Compulsive Scale for Eating Disorders (YBC-EDS)
Description: The YBC-EDS is an eight item, clinician-rated instrument assessing eating related preoccupations and/or rituals. Possible scores range from 0 to 32, with higher scores indicating greater preoccupations. Random effects regression models were used to compare fluoxetine vs placebo groups over time, using data from all patients.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 49 | 44
units on a scale | -0.18 (0.13) | 0.028 (0.13)
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Random effects regression analysis of change during treatment on the YBC-EDS, in fluoxetine vs placebo groups; Test type: Superiority; p = 0.26, Mixed Models Analysis; Reported p values of secondary measures were not corrected for multiple comparisons. The Bonferroni corrected level of significance is <0.005

ADVERSE EVENTS:
Description: Approximately weekly clinician interview over one year
Groups:
- Placebo: Placebo Medication
Arm/Group | Fluoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/44
Other Adverse Events (participants affected / at risk) | 0/49 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=49) | Placebo (N=44)
suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No